CLINICAL TRIAL: NCT07198217
Title: Real World Study of Platinum Containing Dual Drug Chemotherapy Followed by Large Fractionated Radiotherapy Combined withTislelizumab in Stage IIIB/C-IV Non-small Cell Lung Cancer Patient
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zibo Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-Ethical Review -01
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: NSCLC; Tislelizumab; Chemotherapy; Hypofractionated Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: SBRT combined with Tislelizumab followed by Tislelizumab

INTERVENTIONS:
Drug: SBRT combined with Tislelizumab followed by Tislelizumab — The enrolled population consists of patients with stage IIIB/C-IV non-small cell lung cancer who are driver gene negative or unknown, as well as those with driver gene positive targeted drug resistance. The patients reaching SD, PR, or CR after 4 cycles of platinum based dual drug chemotherapy. The patient will receive SBRT radiotherapy combined with Tislelizumab treatment, followed by Tislelizumab maintenance therapy.

SUMMARY:
In clinical practice, some patients cannot tolerate concurrent chemoradiotherapy. The purpose of this study is to observe the efficacy and safety of platinum-based doublet chemotherapy followed by hypofractionated radiotherapy and Tislelizumab in patients with stage IIIB/C-IV non-squamous non-small cell lung cancer. This study aims to provide more treatment options for patients with locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
3. Patients with stage IIIB/C-IV non-squamous non-small cell lung cancer confirmed by cytology or histology;
4. Tumor histology or hematology confirms no EGFR mutations and no mutations or positive driver genes for ALK, BRAF, ROS1, RET, MET, etc or Targeted drug therapy leads to drug resistance progression

Exclusion Criteria:

1. Patients with uncontrolled autoimmune diseases;
2. Patients who have experienced autoimmune reactions within the past 6 months and whose conditions have not improved or are unstable after corresponding treatments, such as pneumonia, thyroiditis, myocarditis, etc. that have not stabilized after treatment;
3. Patients who have previously received systemic chemotherapy, or adjuvant or neoadjuvant therapy, and the time from the last treatment to recurrence is less than 3 months;
4. Patients with known allergies or contraindications to the study drug or its excipients;
5. Pregnant or lactating female patients, or female patients of childbearing potential with a positive baseline pregnancy test;
6. Female patients of childbearing potential or male patients with reproductive plans who are unwilling to use effective contraception during the entire trial period and for 6 months after the end of the trial;
7. Patients whose comorbidities or other conditions may affect compliance with the protocol or are deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
One-year PFS rate | Up to approximately 24 months
  The proportion of patients who survived for more than one year after treatment without disease progression

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS is defined as the time from the first dose until the first documentation of progression or death from any cause, whichever occurs first, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR), as assessed by the investigator using RECIST v1.1.
Overall survival (OS) | Up to ~48 months
  OS is defined as the time from first dose until the date of death due to any cause
Disease Control Rate (DCR) | Up to ~24 months
  DCR is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD), as assessed by the investigator using RECIST v1.1.
Adverse events | Through study completion, an average of 2 year
  The incidence and severity of AEs will be determined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Zibo Municipal Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided